CLINICAL TRIAL: NCT00897949
Title: A Randomized, Triple-Blind, Double-Dummy, Placebo-Controlled, Parallel Groups, Outpatient Study to Examine the Safety and Efficacy of MK0462 10 mg p.o. and MK0462 5 mg p.o. for the Treatment of Acute Migraine and Migraine Recurrence
Brief Title: MK0462 in Treatment of Migraine With Recurrence (MK0462-022)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-022; 2009_589
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2011-05-04 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Rizatriptan 10 mg (Experimental)
  Interventions: Drug: rizatriptan benzoate (MK0462)
- Rizatriptan 5 mg (Experimental)
  Interventions: Drug: rizatriptan benzoate (MK0462)
- Placebo (Placebo Comparator)
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: rizatriptan benzoate (MK0462) — Single dose administration of 5 or 10 mg oral tablet of rizatriptan, taken immediately upon development of acute/severe migraine headache.
  Arms: Rizatriptan 10 mg; Rizatriptan 5 mg
Drug: Comparator: placebo — Placebo to rizatriptan
  Arms: Placebo

SUMMARY:
A study to evaluate rizatriptan/MK0462 (5 and 10 mg) for the treatment of acute migraine attack and treatment of up to two headache recurrences compared to placebo.

The long term extension study which pools patients from MK0462-022, -025, and -029 is described in NCT01286207.

ELIGIBILITY:
Inclusion Criteria:

* Patient had at least a 6-month history of migraine, with or without aura
* Patient was male, or if female must have been postmenopausal, surgically sterilized, or taking adequate contraceptive precautions
* Patient was judged to be in good health, apart from migraine

Exclusion Criteria:

* Patient was pregnant or a nursing mother
* Patient had abused drugs or alcohol within 12 months prior to entering the study
* Patient had a history of cardiovascular disease
* Patient had clinically significant ECG abnormality
* Patient had a resting systolic blood pressure of greater than 145 mm Hg or diastolic of less than 95 mm Hg at screening
* Patient received treatment with an investigational device or compound within 30 days of the study start
* Patient typically suffered from less then 1 or more than 8 attacks of migraine per month
* Patient had difficulty in distinguishing his/her migraine attacks from tension or interval headaches
* Patient had prior exposure to rizatriptan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1473 (Actual)
Dates: Start 1995-03; Primary Completion 1996-01 (Actual); Study Completion 1996-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Ho TW, Rodgers A, Bigal ME. Impact of recent prior opioid use on rizatriptan efficacy. A post hoc pooled analysis. Headache. 2009 Mar;49(3):395-403. doi: 10.1111/j.1526-4610.2009.01346.x. Epub 2008 Feb 12. PMID 19222588
- [Background] Ho TW, Fan X, Rodgers A, Lines CR, Winner P, Shapiro RE. Age effects on placebo response rates in clinical trials of acute agents for migraine: pooled analysis of rizatriptan trials in adults. Cephalalgia. 2009 Jul;29(7):711-8. doi: 10.1111/j.1468-2982.2008.01788.x. Epub 2009 Feb 3. PMID 19210513
- [Result] Teall J, Tuchman M, Cutler N, Gross M, Willoughby E, Smith B, Jiang K, Reines S, Block G. Rizatriptan (MAXALT) for the acute treatment of migraine and migraine recurrence. A placebo-controlled, outpatient study. Rizatriptan 022 Study Group. Headache. 1998 Apr;38(4):281-7. doi: 10.1046/j.1526-4610.1998.3804281.x. PMID 9595867
- [Result] Block GA, Goldstein J, Polis A, Reines SA, Smith ME. Efficacy and safety of rizatriptan versus standard care during long-term treatment for migraine. Rizatriptan Multicenter Study Groups. Headache. 1998 Nov-Dec;38(10):764-71. doi: 10.1046/j.1526-4610.1998.3810764.x. PMID 11284464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 28 sites in the United States and 18 in 9 other countries.
  First Patient Treated: Mar 1995
  Last Patient Treated: Jan 1996.
Pre-assignment Details: Outpatients randomized at the prestudy visit were given study drug and administration instructions. If patients had not treated an attack within 2 months of being enrolled, they were required to return for a rescreen visit. If by 4 months after being enrolled patients still had not treated an attack, they were discontinued from the study
Groups:
- Rizatriptan 5 mg: Rizatriptan 5 mg orally once for treatment of single migraine attack
- Rizatriptan 10 mg: Rizatriptan 10 mg orally once for treatment of single migraine attack
- Placebo: Placebo matching Rizatiptan 5 mg and Rizatriptan 10 mg orally once for treatment
Period: Overall Study
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Placebo
Started | 554 (Patients who were allocated study drug) | 549 (Patients who were allocated study drug) | 370 (Patients who were allocated study drug)
Patients Treated | 458 (Patients who took study drug) | 456 (Patients who took study drug) | 304 (Patients who took study drug)
Completed | 450 (Patients who took study drug and completed the study) | 446 (Patients who took study drug and completed the study) | 301 (Patients who took study drug and completed the study)
Not Completed | 104 | 103 | 69
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Protocol Violation | 6 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Patient Uncoorperative | 0 | 2 | 1
Not completed — Lost to Follow-up | 30 | 23 | 17
Not completed — Withdrawal by Subject | 24 | 31 | 17
Not completed — Abnormal Prestudy Labs | 2 | 3 | 4
Not completed — Abnormal Baseline ECG | 2 | 2 | 4
Not completed — Need for Concom. Med. | 0 | 1 | 1
Not completed — Lack of Migraine Attack | 29 | 30 | 19
Not completed — Did not take study drug | 9 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Placebo | Total
Number analyzed (Participants) | 458 | 456 | 304 | 1218
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (9.6) | 40.7 (9.6) | 40.6 (10.5) | 40.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 394 | 402 | 259 | 1055
  Male | 64 | 54 | 45 | 163
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 430 | 422 | 286 | 1138
  Black | 18 | 7 | 7 | 32
  Asian | 2 | 12 | 3 | 17
  Hispanic | 0 | 1 | 1 | 2
  Mexican-American | 0 | 1 | 0 | 1
  Syrian | 0 | 0 | 1 | 1
  Anglo-Asian | 1 | 0 | 0 | 1
  Mixed | 3 | 4 | 1 | 8
  Other | 4 | 9 | 5 | 18
Baseline Headache Severity [Number; unit: Participants] — Each patient rated headache severity on a 4-grade scale (0 = no headache; 1 = mild pain; 2 = moderate pain; 3 = severe pain)
  Participants
    Grade 0, 1: No pain, Mild, or missing | 8 | 9 | 7 | 24
    Grade 2: Moderate | 298 | 316 | 202 | 816
    Grade 3: Severe | 152 | 131 | 95 | 378

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief at 2 Hours After the Initial Dose of Test Drug
Description: Patients reporting pain relief (defined as a reduction of headache severity from grades 2/3 at baseline to 0/1) at 2 hours after the initial dose of test drug. Pain severity was subjectively rated by patients on a scale from grade 0 to 3: Grade 0 - No headache, Grade 1 - Mild pain, Grade 2 - Moderate pain, Grade 3 - Severe pain.
Time Frame: 2 hours after initial dose of test drug
Population: The primary analysis employed an "all-patients-treated" approach that included all patients who had at least one record of pain severity within 2 hours after the initial dose. Missing data were replaced by carrying forward the preceding value.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 457 | 455 | 302
Participants
  Reporting pain relief | 285 | 322 | 106
  Not reporting pain relief | 172 | 133 | 196

2. Secondary Outcome: Pain Free at 2 Hours After the Initial Dose of Test Drug
Description: Patients reporting pain free (defined as a reduction of headache severity to grade 0 [no pain]) at 2 hours after the initial dose of test drug. Pain severity was subjectively rated by patients on a scale from grade 0 to 3: Grade 0 - No headache, Grade 1 - Mild pain, Grade 2 - Moderate pain, Grade 3 - Severe pain.
Time Frame: 2 hours after initial dose of test drug
Population: An "all-patients-treated" approach was employed that included all patients who had at least one record of pain severity within 2 hours after the initial dose. Missing data were replaced by carrying forward the preceding value.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 457 | 455 | 302
Participants
  Reporting no pain | 150 | 193 | 30
  Reporting pain | 307 | 262 | 272

3. Secondary Outcome: No Disability at 2 Hours After the Initial Dose of Test Drug
Description: Patients with no disability at 2 hours after the initial dose of test drug. Functional disability was subjectively rated on a scale from grade 0 to 3: Grade 0 - Normal, Grade 1 - Daily activities mildly impaired, Grade 2 - Daily activities severely impaired, Grade 3 - Unable to carry out daily activities, requires bedrest
Time Frame: 2 hours after initial dose of test drug
Population: An "all-patients-treated" approach was employed that included all patients who had at least one record of functional disability within 2 hours after the initial dose. Missing data were replaced by carrying forward the preceding value.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 457 | 454 | 300
Participants
  Normal | 175 | 209 | 54
  Mildly Impaired | 160 | 148 | 118
  Severely Impaired | 56 | 45 | 53
  Requires Bedrest | 66 | 52 | 75

4. Secondary Outcome: Use of Escape Medication at 2 Hours After the Initial Dose of Test Drug
Time Frame: 2 hours after initial dose of test drug
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 458 | 456 | 304
Participants
  Used escape medication | 101 | 76 | 128
  Did not use escape medication | 357 | 380 | 176

5. Secondary Outcome: Pain Relief 2 Hours After Treatment for Headache Recurrence
Description: Patients reporting pain relief 2 hours after treatment for headache recurrence (defined as the return of headache to grade 2 or 3 within 24 hours of the initial dose in patients who reported pain relief (grades 0 or 1) at 2 hours).
Time Frame: 2 hours after treatment for recurrence
Population: Patients with initial headache recurrence who took rizatriptan 5 mg or 10 mg were prerandomized (ratio=1:1) to either rizatriptan 5 mg or 10 mg, respectively, or to placebo (ratio=1:1); and who took placebo, to either 5 mg or 10 mg of rizatriptan (ratio=1:1). Only those who took rizatriptan for their initial headache were considered for analysis.
Measure: Number; unit: Participants
Groups:
- Rizatriptan 5 mg / Rizatriptan 5 mg: Rizatriptan 5 mg initially, prerandomized to rizatriptan 5 mg
- Rizatriptan 5 mg / Placebo: Rizatriptan 5 mg initially, prerandomized to placebo
- Rizatriptan 10 mg / Rizatriptan 10 mg: Rizatriptan 10 mg initially, prerandomized to rizatriptan 10 mg
- Rizatriptan 10 mg / Placebo: Rizatriptan 10 mg initially, prerandomized to placebo
- Placebo / Rizatriptan 5 mg: Placebo initially, prerandomized to rizatriptan 5 mg
- Placebo / Rizatriptan 10 mg: Placebo initially, prerandomized to rizatriptan 10 mg
Arm/Group | Rizatriptan 5 mg / Rizatriptan 5 mg | Rizatriptan 5 mg / Placebo | Rizatriptan 10 mg / Rizatriptan 10 mg | Rizatriptan 10 mg / Placebo | Placebo / Rizatriptan 5 mg | Placebo / Rizatriptan 10 mg
Number analyzed (Participants) | 55 | 59 | 65 | 75 | 17 | 22
Participants
  Pain relief | 39 | 32 | 53 | 33 | 12 | 18
  No pain relief | 16 | 27 | 12 | 42 | 5 | 4

ADVERSE EVENTS:
Time Frame: During the 24 hours treatment period, and up to and including 7 days after the last dose of study therapy.
Description: Although a patient may have had two or more adverse experiences the patient is counted only once in a category. The same patient may appear in different categories.
  The subjects reported at risk are subjects with follow-up after at least one dose of study drug.
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/456 | 0/455 | 0/307
Other Adverse Events (participants affected / at risk) | 155/456 | 254/455 | 83/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan 5 mg (N=456) | Rizatriptan 10 mg (N=455) | Placebo (N=307)
Headache (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan 5 mg (N=456) | Rizatriptan 10 mg (N=455) | Placebo (N=307)
Asthenia/Fatigue (General disorders) | 12 | 33 | 6
Pain, Abdominal (General disorders) | 6 | 9 | 4
Pain, Chest (General disorders) | 7 | 12 | 2
Dry Mouth (Gastrointestinal disorders) | 11 | 15 | 5
Nausea (Gastrointestinal disorders) | 19 | 22 | 14
Vomiting (Gastrointestinal disorders) | 9 | 10 | 4
Alanine Amino Transferase (ALT) Increased (Investigations) | 3 | 3 | 2
Aspartate Amino Transferase (AST) Increased (Investigations) | 1 | 3 | 2
Tightness, Regional (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0
Disorientation (Nervous system disorders) | 0 | 5 | 0
Dizziness (Nervous system disorders) | 19 | 45 | 14
Headache (Nervous system disorders) | 7 | 8 | 2
Hypesthesia (Nervous system disorders) | 4 | 4 | 4
Insomnia (Nervous system disorders) | 5 | 2 | 0
Paresthesia (Nervous system disorders) | 11 | 17 | 4
Somnolence (Nervous system disorders) | 16 | 37 | 9
Tremor (Nervous system disorders) | 6 | 1 | 5
Discomfort, Pharyngeal (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 0
Infection, Respiratory, Upper (Infections and infestations) | 5 | 4 | 1
Flushing (Skin and subcutaneous tissue disorders) | 4 | 4 | 4
Hot Flashes (Reproductive system and breast disorders) | 2 | 5 | 1

LIMITATIONS AND CAVEATS:
Pooled Extension data for PN022- NCT00897949; PN025- NCT00899379 and PN029- NCT00897104 appears in NCT01286207

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.